CLINICAL TRIAL: NCT01733355
Title: A Phase 0, Open Label, Non-randomized, Multi-center Exploratory and Safety Study of [F-18]T807
Brief Title: A Phase 0, Open Label, Multi-center Exploratory and Safety Study of [F-18]T807
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study was terminated in anticipation of transfer of ownership to Avid Radiopharmaceuticals.
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: T807000
Record Dates: First submitted 2012-09-25; First posted 2012-11-27 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Alzheimers Disease; AD
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole; tau Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tau diagnostic (Experimental): [F18] T807
  Interventions: Radiation: [F18] T807

INTERVENTIONS:
Radiation: [F18] T807 — Dose for normal volunteer undergoing dosimetry evaluation will not exceed 20 mCi, dose for high probability of Alzheimer's and low probability Alzheimer's undergoing brain imaging only will not exceed 10 mCi
  Other Names: Tau [F-18]T807

SUMMARY:
[F-18]T807 is being developed as a diagnostic radiopharmaceutical for PET imaging of the human brain.

DETAILED DESCRIPTION:
Siemens Molecular Imaging (SMI) is seeking to determine if [F-18]T807 might be useful as a non-invasive assessment tool in the clinical evaluation of subjects with conditions associated with tau protein aggregates, such as Alzheimer's disease. The information collected under this exploratory study will not be used for diagnostic purposes, assessments of the participant's response to therapy or for clinical management of the participants. However, this exploratory study will provide baseline information on the safety, biodistribution, and dosimetry of [F-18]T807. These data will aid in the design of future studies of [F-18]T807 in patients with Alzheimer's disease. Overall, this study will provide initial data that inform the development of [F-18]T807 as the first PET imaging agent for human tau protein related pathology.

ELIGIBILITY:
Inclusion Criteria; Low Probability for AD Participants (Group 1)

* Participant has reached his or her 55th birthday at the time of informed consent (Participant is male or female of any race / ethnicity)
* Participant provides written informed consent
* Participant is capable of complying with study procedures
* Participant is capable of communicating with study personnel
* Participant understands and speaks English
* Participant has at least an 8th Grade education
* In the Investigator's opinion, participant has a low probability of being currently positive for AD as determined by a Mini Mental State Examination (MMSE ≥ 28) defined in APPENDIX VI of protocol T807000, IND 114102
* Participant has no significant hepatic or renal disease as defined by previous medical history and lab results are within the following ranges:
* Total bilirubin within 2x institutional upper limits of normal
* AST (SGOT) ≤ 2.5 x institutional upper limits of normal
* ALT (SGPT) ≤ 2.5 x institutional upper limits of normal
* Creatinine ≤ 2x institutional upper limits of normal
* BUN within 2x institutional upper limits of normal

High Probability for AD Participants (Group 2)

* Participant has reached his or her 55th birthday at the time of informed consent (Participant is male or female of any race / ethnicity)
* Participant or participant's legally acceptable representative provides written informed consent
* Participant is capable of complying with study procedures
* Participant is capable of communicating with study personnel
* Participant understands and speaks English
* Participant has at least an 8th Grade education
* In the Investigator's opinion, participant has a high probability of being currently positive for AD that is determined by a Mini Mental State Examination (MMSE < 17) defined in APPENDIX VI of protocol T807000, IND 114102.
* Participant has no significant hepatic or renal disease as defined by previous medical history, and lab results are within the following ranges:
* Total bilirubin within 2x institutional upper limits of normal
* AST (SGOT) ≤ 2.5 x institutional upper limits of normal
* ALT (SGPT) ≤ 2.5 x institutional upper limits of normal
* Creatinine ≤ 2x institutional upper limits of normal
* BUN within 2x institutional upper limits of normal

Exclusion Criteria; All Participants

* Female participant is pregnant or nursing
* Participant has prior history of stroke or other condition of the head or neck that, in the Investigator's opinion, might affect circulation to the head or image interpretation
* Participant has other neurodegenerative disease that is associated with cognitive impairment or dementia
* Participant has a medical condition that might be associated with elevated amyloid levels, such as amyloid angiopathy, familial amyloidosis, chronic kidney dialysis, Down's syndrome
* Participant has a history of significant cerebrovascular disease
* Participant has previously received [F-18]T807 at any time
* Participant has been involved in an investigative, radioactive research procedure within the past 14 days
* Participant has any other condition or personal circumstance that, in the judgment of the Investigator, might interfere with the collection of complete data or data quality
* Participant has a history in the last five years of significant prescription or non-prescription drug or alcohol abuse, including but not limited to marijuana, cocaine, heroin or derivatives

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the bio-distribution and radiation dosimetry of [F-18]T807 in participants with low probability of Alzheimer's disease (AD) using PET/CT whole body imaging | up to 15 days per patient
To evaluate the metabolism of [F-18]T807 in participants with low probability of AD using serial blood samples collected pre- and post-IP administration | up to 15 days per patient
To evaluate [F-18]T807 uptake and signal/background information in brain PET/CT imaging of participants with a high probability of currently being positive for AD and age-matched participants with a low probability of currently being positive for AD | upto 15 days per patient
To assess the safety of IV administration of [F-18]T807 | up to 24 hours post [F18]T807 administration
  Safety will be monitored for all subjects by the:
  * Number of subjects experiencing adverse events from baseline to 24 hours post-administration.
  * Number and type of adverse events.
  * Changes in clinical laboratory assessments (CBC and clinical chemistry)from baseline to 24 hours post administration.
  * Changes in physical examination from baseline to 24 hours post administration.
  * Changes in vital sign measurements (systolic blood pressure [mmHg]; diastolic blood pressure [mmHg], pulse rate [bpm] and body temperature) from baseline prior to [F-18]T807 administration, at 60 +/- 15 minutes post administration, at the end of the final imaging session (approximately 100 minutes post administration)and at 24 hours post administration.
  * Changes in ECG measurements, from baseline prior to [F-18]T807 administration, at 60 +/- 15 minutes post administration, at the end of the final imaging session (approximately 100 minutes post administration) and at 24 hours post administration.

SECONDARY OUTCOMES:
To begin collection of baseline [F-18]T807 PET/CT imaging data | up to 15 days per patient
  The secondary endpoint of this investigational study is the collection of baseline whole body PET/CT images and PET/CT images of the brain, following administration of [F-18]T807
To gain information to improve the study design for the conduct of future trials | up to 15 days per patient
  The secondary endpoint of this investigational study is the collection of baseline whole body PET/CT images and PET/CT images of the brain, following administration of [F-18]T807

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (2):
- United States (2):
  - Research Site, Irvine, California
  - Research Site, Los Angeles, California